CLINICAL TRIAL: NCT02405728
Title: Vascular Access in Hematological Patients - PICC Versus CVC in a Phase IV Randomized Controlled Trial
Brief Title: Vascular Access in Hematological Patients - PICC Versus CVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Prof, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HEM-FEDII-PICC-001
Record Dates: First submitted 2015-03-13; First posted 2015-04-01 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Vascular Access Complication
Keywords: PICC; BLOODSTREAM INFECTIONS; VASCULAR ACCESS; DEEP VEIN THROMBOSIS; CICC
MeSH Terms: conditions — Sepsis; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripherally inserted central catheters (Experimental): Peripherally inserted central catheters (PICCs) - Most commonly used vascular access in hematological patients - Randomization between CICCs and PICCs
  Interventions: Device: Peripherally inserted central catheters (PICCs)
- Centrally inserted central catheter (Active Comparator): Centrally inserted central catheter (CICCs) - New vascular access, with the aim to reduce the complications - Randomization between CICCs and PICCs
  Interventions: Device: Centrally inserted central catheters (CICCs)

INTERVENTIONS:
Device: Centrally inserted central catheters (CICCs) — Randomization between two well established clinical routine vascular access devices
  Arms: Centrally inserted central catheter
Device: Peripherally inserted central catheters (PICCs) — Randomization between two well established clinical routine vascular access devices
  Arms: Peripherally inserted central catheters

SUMMARY:
The use of peripherally inserted central catheters (PICCs) represents a major advance for hematological patients, enabling the effective delivery of chemotherapy and/or blood products particularly for prolonged infusions or in situation of difficult venous access. In modern medical practice their use has increased rapidly for several reasons, including ease of insertion, many uses (e.g., drug administration and venous access), perceived safety, and cost-effectiveness compared with centrally inserted central catheters (CICCs).

DETAILED DESCRIPTION:
The use of peripherally inserted central catheters (PICCs) represents a major advance for hematological patients, enabling the effective delivery of chemotherapy and/or blood products particularly for prolonged infusions or in situation of difficult venous access. In modern medical practice their use has increased rapidly for several reasons, including ease of insertion, many uses (e.g., drug administration and venous access), perceived safety, and costeffectiveness compared with centrally inserted central catheters (CICCs). Despite these benefits, PICCs are associated with deep vein thrombosis of the arm and pulmonary embolism. These complications, which are often called venous thromboembolism, are important because they not only complicate and interrupt treatment, but also increase cost, morbidity and mortality. Despite this effect, the burden and risk of PICC-related venous thromboembolism is uncertain and clinicians have scarce evidence on which to base choice of vascular access. Evidence to choose one vascular access over the other is lacking in literature, in particular for patients affected by haematological malignancies, in which chemotherapy is more likely to cause myelosuppression, with a major risk of bloodstream infections. Furthermore, the precise incidence and the risk of PICC-related venous thromboembolism relative to that of other CICCs is unknown. An understanding of this risk in the context of growing PICC use is an important cost and patients safety questions. Up to now, no systematic review has been done to investigate these questions.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yrs
* Newly diagnosed AML
* Suspected survival > 4 weeks
* Need of central venous access >4 weeks

Exclusion Criteria:

* Ongoing uncontrolled systemic infection
* Presence of significant thrombosis/stenosis in arm or central veins
* Diagnosis of another cancer within 12 months before AML onset
* any evidence of clinical conditions indicating unability to receive intent-to- cure chemotherapy
* Unability to communicate and/or to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Catheter-related bloodstream infections | 1 year
  1. Cumulative incidence of catheter-related (CR)-major complications: catheter-related bloodstream infections and CR-deep-vein thrombosis.

SECONDARY OUTCOMES:
Other complications | 1 year
  2. Occurrence of complications associated with catheter positioning (serious bleeding, arterial puncture and/or pneumothorax), catheter malfunctions (dislocation, occlusion and/or rupture), catheter removals and 30-days overall mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Picardi, Prof, Principal Investigator — Hematology - AOU Federico II - Napoli - Italy
Locations (1):
- Prof Marco Picardi - Hematology - AOU FEDERICO II, Napoli, Italy